CLINICAL TRIAL: NCT05422521
Title: Radiomics and Metabolomics in the Follow-up of CAR T-cells for Refractory or Relapsed Non-Hodgkin's Lymphoma: Pilot Study
Brief Title: Radiomics and Metabolomics in the Follow-up of CAR T-cells for Refractory or Relapsed Non-Hodgkin's Lymphoma
Acronym: CART-Omic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-AOIP-03
Record Dates: First submitted 2022-05-31; First posted 2022-06-16 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Refractory or Relapsed Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- identification of predictive and prognostic biomarkers (Experimental)
  Interventions: Other: blood samples and 18FDG PET-CT exams

INTERVENTIONS:
Other: blood samples and 18FDG PET-CT exams — * 18 FDG PET scanner at inclusion and post CART-cells treatment ( 1, 3, 6, 9 and 12 month)
  * blood collection at inclusion and post CART-cells treatment (7 days, 1 month and 3 month)

SUMMARY:
This is an interventionnal pilot study to investigate whether 18FDG radiomics or serum metabolomic signatures could be predictive or prognostic factors in the follow-up of patients receiving CAR T-cell therapy for refractory non-Hodgkin's lymphoma or in relapse.

DETAILED DESCRIPTION:
In this study the search for relevant radiomic signature will be carried out for each patient benefiting from an 18FDG PET-CT during the pre-treatment assessment and then in the follow-up at 1 month, 3 months, 6 months, 9 months and 12 months post treatment.

The search for circulating metabolites in serum (mass spectrometry) will be carried out during the pre-therapeutic assessment, then in the follow-up at 7 days, 1 month, 3 months, 6 months, 9 months and 12 months post treatment.

The main objective of the study is the comparison of signatures from radiomics and early serum metabolomic indices according to progression-free survival at 12 months of patients treated with CAR T-cells for refractory or relapsed non-Hodgkin's lymphoma, in correlation with clinical and biological monitoring, to predict tumor response.

The secondary objective is the comparison of the signatures of early serum radiomic and metabolic indices according to the occurrence of serious clinical and/or biological side effects in the 12 months following treatment with CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Patients with histologically proven, refractory or relapsed, non-Hodgkin's lymphoma as indicated for CAR T-cell therapy
* ECOG score 0 to 2
* Affiliated patient or beneficiary of a social security scheme
* Patient having signed prior informed consent.

Exclusion Criteria:

* Be under 18 years old,
* Contraindication to performing 18FDG PET-CT examinations: severe claustrophobia, unbalanced diabetes during PET-CT examinations (young capillary blood sugar ≥ 11 mmol),
* Any participation in other biomedical studies relating to drugs, medical devices or imaging techniques is prohibited, with the exception of so-called non-health product biomedical studies.
* Hypersensitivity to the active substance or to any of the excipients in the composition of CAR T-cells preparations
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) compared and correlated with signatures of the radiomics and serum metabolomics index | 7 days, 1 month, 3 months, 6 months, 9 months and 12 months post treatment.
  Progression-free survival (PFS)

SECONDARY OUTCOMES:
Occurrence of severe side effects compared and correlated with the signatures of the radiomics and serum metabolomics indexes. | 7 days, 1 month, 3 months, 6 months, 9 months and 12 months after injection
  occurrence of severe side effects

CONTACTS AND LOCATIONS:
Overall Officials: Philippe VIAU, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No